CLINICAL TRIAL: NCT02763813
Title: Comparison of a Retention Type and Propulsion Type Oral Appliance in the Treatment of Obstructive Sleep Apnea
Brief Title: Comparison of Two Oral Appliances in the Treatment of Sleep Apnea Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/05
Record Dates: First submitted 2016-04-19; First posted 2016-05-05 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propulsion type appliance (Herbst) (Experimental)
  Interventions: Device: Herbst (propulsion type oral appliance)
- Retention type appliance (ORM) (Active Comparator): Retention type appliance
  Interventions: Device: Retention type appliance (ORM)

INTERVENTIONS:
Device: Herbst (propulsion type oral appliance) — Oral appliance
  Arms: Propulsion type appliance (Herbst)
Device: Retention type appliance (ORM)
  Arms: Retention type appliance (ORM)

SUMMARY:
Monocentric comparative group study comparing the efficacy and short-term tolerance of a propulsion type oral appliance (Herbst) with a retention type device (ORM) used in the treatment of sleep apnea syndrome. The investigators hypothesized both appliances would be equally effective and tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient teeth to allow wearing of the device
* Mild to severe OSAS
* Ability to answer the questionnaires
* No concomitant CPAP treatment
* BMI inferior to 32 kg/m2

Exclusion Criteria:

* Important dental or parodontal disease
* Central sleep apnea
* Jaw opening limitations
* Temporo-mandibular joint dysfunction
* Major gag reflex precluding the long-term use of the device
* Major or unstable cardiovascular or pulmonary disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Apnea/hypopnea index (as measured from a level 1 or 2 polysomnography) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc BLUMEN, MD, Study Chair — Hôpital FOCH 40, rue Worth 92150 Suresnes
Locations (1):
- Hôpital FOCH, Suresnes, France